CLINICAL TRIAL: NCT07368699
Title: Evaluation of Active Oxygen Releasing Gel Combined With Photodynamic Therapy in The Treatment of Stage III Periodontitis (A Randomized Controlled Clinical Trial)
Brief Title: Active Oxygen Releasing Gel With Photodynamic Therapy in Treating Stage III Periodontitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Aya Abdelmawla, Periodontology resident at periodontology department Alexandria University,Egypt, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1016-12/2024
Record Dates: First submitted 2026-01-17; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Stage III Periodontitis
Keywords: Active oxygen releasing gel; Photodynamic therapy; Periodontitis; Scaling and Root Planing,
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Masking Description: The study is open-label for participants and clinicians due to the nature of the interventions. However, to ensure objectivity, the trial statistician and the microbiologist performing the laboratory analysis will remain masked to treatment assignment (blinded) until the final data analysis is complete. Samples sent to the microbiology lab will be coded with unique identification numbers to maintain blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SRP+Active oxygen gel. (Experimental): Scaling and root planing(SRP)followed by topical application of active oxygen-releasing gel (0.4 mL) for 3 minute
  Interventions: Procedure: Scaling and root planing and topical application of active oxygen-releasing gel; Procedure: Scaling and root planing
- SRP+ Oxygen gel+Laser (Experimental): Scaling and root planing (SRP) will be performed in a single session, followed by the topical application of active oxygen-releasing gel (0.4 mL) for 3 minutes. Subsequently, antimicrobial Photodynamic Therapy (aPDT) will be applied using a diode laser (635 nm) with tolonium chloride as a photosensitizer. The laser irradiation will be performed at an energy density of 6 J/cm2 for 30 seconds per site."
  Interventions: Procedure: Scaling and root planing, topical active oxygen-releasing gel, and photodynamic therapy using diode laser; Procedure: Scaling and root planing and topical application of active oxygen-releasing gel; Procedure: Scaling and root planing
- Scaling and root planing alone. (Active Comparator): Scaling and root planing using ultrasonics and Gracey curettes.
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Procedure: Scaling and root planing, topical active oxygen-releasing gel, and photodynamic therapy using diode laser — 14 stage III periodontitis patients will undergo scaling and root planing in a single session followed by topical application of active oxygen-releasing gel (0.4 mL) for 3 minutes then irrigating the targeted pocket using tolonium chloride will be stopped once the tolonium chloride solution will be observed at the free gingival margin of the pocket. After 60 seconds, irradiation inside the periodontal pocket with diode laser (635nm) for 200 mW, 30 seconds, energy density of 6 J/cm2, tip diameter of 400 µm, using continuous modes of irradiation, the laser fiber tip will be positioned parallel to the long axis of the tooth, move in a steady vertical inward and outward motion to ensure that the entire pocket will be adequately covered.
  Arms: SRP+ Oxygen gel+Laser
Procedure: Scaling and root planing and topical application of active oxygen-releasing gel — 14 patients with stage III periodontitis will undergo scaling and root planing in a single session followed by topical application of active oxygen-releasing gel (0.4 mL) for 3 minutes.
  Arms: SRP+ Oxygen gel+Laser; SRP+Active oxygen gel.
Procedure: Scaling and root planing — 14 patients will undergo scaling and root planing(SRP) using ultrasonics and Gracey curettes.

SUMMARY:
Periodontitis is a serious gum disease that can damage the tissues supporting the teeth. The standard treatment is scaling and root planing of the teeth and roots. However, in some patients, this treatment alone may not fully control inflammation and harmful bacteria.

This study aims to evaluate whether adding an active oxygen-releasing gel, with or without photodynamic therapy, improves treatment outcomes in patients with stage III periodontitis. The oxygen-releasing gel is applied to the gums and releases oxygen, which may help reduce harmful bacteria. Photodynamic therapy uses a light source together with a special dye to target and destroy bacteria and improve gingival health.

In this randomized clinical trial, 42 patients with stage III periodontitis will be divided into three groups. One group will receive standard scaling and root planing (SRP) plus the oxygen-releasing gel. A second group will receive standard scaling and root planing (SRP)plus the gel and photodynamic therapy. The third group will receive standard scaling and root planing(SRP) only.

Gum health will be evaluated by measuring gingival index, bleeding index, pocket depth, and supra crestal tissue attachment level at the start of the study and after one and three months. Microbiological samples from periodontal pockets will also be used to assess levels using quantitative Polymerase Chain Reaction (qPCR) for relative abundance of Treponema denticola and Porphyromonas gingivalis bacteria related to periodontal disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with periodontal diagnosis of stage III periodontitis
* Patients with residual periodontal pocket depth ≥4 mm ,CAL≥ 5mm with bone loss extending to middle third of root and beyond in radiography
* Bleeding on probing at least four sites at base-line
* Patients who didn't receive periodontal treatment for a minimum of 3 months prior to the examination.
* Patients of both sexes aged ≥30 and ≤70 years

Exclusion Criteria:

* Smokers or those with any other harmful habits such as pipe or vape smoking
* Patients with any systemic condition that will possibly affect the outcome of periodontal therapy i.e. (diabetic patients)
* Patients who have received any local or systemic anti-inflammatory medications or antibiotics within the last 6 months
* Pregnant or lactating women
* Patients with parafunctional habits

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-01-26 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Modified Gingival Index (MGI) score | Before enrollment, and one and three months after enrollment
  non-invasive, visual clinical tool (0-4 scale)focuses on color, texture, and contour changes across facial, lingual, mesial, and distal surfaces of tooth ,modified gingival Scoring Criteria for MGI (0-4) higher scores indicate more severe gingival inflammation higher a worse clinical outcome.
  0: Absence of inflammation (normal gingiva).
  1. Mild inflammation - slight change in color/texture in part of the marginal or papillary gingiva.
  2. Mild inflammation - slight change in color/texture in the entire marginal or papillary gingiva.
  3. Moderate inflammation - bright surface, erythema, edema, and/or hypertrophy of the marginal or papillary gingiva.
  4. Severe inflammation - severe erythema, edema, and/or marg
Percentage of sites with Bleeding on Probing (BOP) assessed by a periodontal probe | Before enrollment, and one and three months after enrollment
  a clinical parameter measured by inserting a periodontal probe to the base of a gingival pocket.The probe is inserted parallel to the root surface and "walked" around the gingival sulcus, with bleeding assessed 30-60 seconds after probing.recorded as a percentage of positive bleeding sites out of the total sites probed (6 sites per tooth). A higher percentage of bleeding sites indicates increased gingival inflammation and a worse outcome.
Measurement of Clinical Attachment Level (CAL) using a Williams calibrated periodontal probe | Before enrollment, and one and three months after enrollment
  measured in millimeters using Williams calibrated probe from the cemento-enamel junction to the bottom of the pocket .This measure reflects the extent of periodontal tissue destruction. Higher values in millimeters indicate greater attachment loss and a worse clinical condition.
Probing Pocket Depth (PPD) in millimeters measured by Williams periodontal probe | Before enrollment, and one and three months after enrollment
  Clinical measurement of the distance in millimeter from the gingival margin to the base of the periodontal pocket using Williams calibrated probe.Deeper pockets indicate more severe periodontal disease. Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Relative abundance of Treponema denticola and Porphyromonas gingivalis using quantitative Polymerase Chain Reaction (qPCR) | Before enrollment and one month after enrollment
  Sub-gingival dental plaque biofilm (before the intervention and one month after the intervention) will be collected using size 30 paper point after ensuring good isolation of the operating field. quantitative real time PCR will be performed using universal bacterial 16SrRNA gene primers and species-specific primers targeting the 16S rRNA genes of Treponema denticola (Td), and Porphyromonas gingivalis (Pg), to estimate the relative abundance of Td and Pg among total oral microbiota before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mohey eldin Elrashidy, PhD,prof, Principal Investigator — Faculty of Dentistry periodontology department Alexandria University,Egypt.; Tarek Alsahry, Phd, Study Director — Faculty of Dentistry periodontology department Alexandria University,Egypt.; Aliaa Gamaleldin Aboulela, PhD, Study Director — Microbiology Department ,Medical Research Institute Alexandria University,Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Bab Sharq, Egypt

IPD SHARING:
Plan to Share IPD: No